CLINICAL TRIAL: NCT02374294
Title: A Prospective, Randomized, Parallel Study Comparing Transdermal, Continuous Oxygen Therapy (TCOT) to Standard of Care to Assess Postoperative Wound Infection Rate in Perineal Resections
Brief Title: TCOT Effectiveness in Preventing Wound Infections in Perineal Resections
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: could not come to budget agreement
Sponsor: Neogenix, LLC dba Ogenix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EPF-614
Record Dates: First submitted 2015-02-11; First posted 2015-02-27 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Complication of Surgical Procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epiflo (Experimental): After the surgery, but before the application of dressing to the surgical site the kit containing the investigation device (and four cannula) is opened. The EPIFLO cannula (sterile package) is opened and applied to the surgical site and sealed with the dressings per protocol. The EPIFLO device is connected to the cannula after making sure the switch is in the ON position.The EPIFLO device is mounted on the patient's body in a convenient location using the Pouch and Arm band provided. At Treatment Visit 3 (Postoperative day #14, +/- 1 day) a new device is given and the old one disposed of. Intermittent dressing changes will take place as needed.
  Interventions: Device: Epiflo
- Standard of Care (No Intervention): After the surgery, but before the application of dressing to the surgical site if upon opening, the kit contains only a weighted block, then, the regular wound dressing protocol, standard of care, will be followed. Intermittent dressing changes will take place as needed.

INTERVENTIONS:
Device: Epiflo — EPIFLO: Small, silent disposable, battery-operated oxygen concentrator capable of delivering 98% to 100% oxygen (balance moisture) for seven days at a rate of ~3.0 ml/hour; and 60" long sterile cannula (tube) that conveys the oxygen concentrator to the area beneath the bandage overlying the wound.
  Arms: Epiflo

SUMMARY:
In colorectal surgery, oxygen insufflation (which leads to higher oxygen concentration in the surgical site) has been shown to decrease infection rate. Several pressure wounds in the coccyx have been successfully treated to closure with Transdermal Continuous Oxygen Therapy (TCOT) Given the wound healing properties of TCOT, particularly in infection-prone anatomic locations such as coccyx, and the microbicidal properties of oxygen, it is expected that the infection rate in abdominoperineal (AP) resection surgery can be reduced with transdermal continuous oxygen therapy. The primary objective of this study is to compare the number of surgical site infections associated with perineal surgery within 28 days between subjects randomized to receive EPIFLO or Standard of Care

DETAILED DESCRIPTION:
EPIFLO is a Small, silent disposable, battery-operated oxygen concentrator capable of delivering 98% to 100% oxygen (balance moisture) for seven days at a rate of ~3.0 ml/hour; and 60" long sterile cannula (tube) that conveys the oxygen concentrator to the area beneath the bandage overlying the wound.

The primary objective of this study is to compare the number of surgical site infections associated with perineal surgery within 30 days between subjects randomized to receive EPIFLO or Standard of Care. Secondary Study objectives include Resource utilization and duration of hospitalization.

Hypothesis 1: The proportion of surgical site infections will be lower for patients treated with Transdermal Continuous Oxygen Therapy (TCOT) Hypothesis 2: In the patients who develop infections, wounds will be smaller and heal more rapidly in those treated with Transdermal Continuous Oxygen Therapy.

Key Safety Assessments Include potential dermatological toxicity changes attributed to EPIFLO as measured by observed and reported discomfort and changes in skin during and after the Treatment Period (It is essential to establish the difference between toxicity from the dressing vs. toxicity arising out of EPIFLO).

This Study will be a randomized controlled trial of 30 patients aged 18-80 years who are scheduled to undergo elective perineal resection surgery at the University of Maryland Medical Center. This study is designed to be a Phase II safety & efficacy study. Patients who met the inclusion/exclusion criteria will be randomized to receive the interventional device with Standard of Care or Standard of Care only (1:1). The patients will be equally divided between the two arms. Sham devices are not involved in this study. Wound infections will be diagnosed by the investigator using Centers for Disease Control and Prevention Criteria. As an additional measure to prevent bias, the pictures of the wounds may be sent to an independent clinical specialist for assessment of infection; this specialist will be blinded to get an objective opinion.

The expected time on study is 1 month ( 27-30 days). This does not include screening period which occurs when the subject consents to be in the study (signs the informed consent) to when they have their surgery (day 1). The screening period can be up to 28 days. While in the study, there are four study visits: Visit 1 day 1 is the day of the surgery, and randomization. The second study visit will be the day of the post surgery discharge (day 3-5). The third study visit will be 14 days following surgery, (day 14) and the Final study visit will be the day of the post surgical follow up visit (day 28). The total treatment period may be 14 or 28 days. After 14-days of treatment, if the wound is completely healed, the treatment phase is complete. If the wound is not completely healed they will receive an additional 14 days of treatment. Either way the patient's healing progress will be followed for a total study duration of 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Elective perineal resection,
* Patients having abdominal-perineal resections or perineal resections will be included.
* Patient age: 18-80

Exclusion Criteria:

* • expected surgery time of less than one hour,

  * fever or existing signs of infection at the time of surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
number of surgical site infections | 30 days
  number of surgical site infections associated with perineal surgery within 30 days between subjects randomized to receive EPIFLO or Standard of Care.

SECONDARY OUTCOMES:
resource utilization (duration of time in hospital) | 30 days